CLINICAL TRIAL: NCT05359445
Title: A Phase Ia/Ib First-In-Human Clinical Trial to Evaluate the Safety, Tolerability and Initial Anti-Tumor Activity of IMA401, a Bispecific T Cell Engaging Receptor Molecule (TCER®), as Monotherapy or in Combination With Checkpoint Inhibitor in Patients With Recurrent and/or Refractory Solid Tumors.
Brief Title: IMA401 TCER® in Recurrent and/or Refractory Solid Tumors, Alone or in Combination With a Checkpoint Inhibitor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA401-101; 2023-506854-19-00 (Other: Clinical Trials Information System)
Record Dates: First submitted 2022-04-11; First posted 2022-05-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Refractory Cancer; Recurrent Cancer; Solid Tumor, Adult; Cancer
Keywords: MAGE-A4
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose-Finding IMA401 TCER® Monotherapy (Phase Ia) (Experimental): Dose-Finding Escalation/De-escalation with IMA401 TCER® (Phase Ia)
  Interventions: Biological: IMA401 (Phase Ia)
- Dose-Finding Combination Therapy with IMA401 TCER® and Pembrolizumab (Phase Ia) (Experimental): Dose-Finding Escalation/De-escalation of combination therapy with IMA401 TCER and pembrolizumab (Phase Ia)
  Interventions: Biological: IMA401 (Phase Ia); Biological: Pembrolizumab (Phase Ia)
- Extension IMA401 TCER® Monotherapy (Phase Ib) (Experimental): IMA401 monotherapy extension cohort following the determination of the recommended dose for extension (RDE) (Phase Ib)
  Interventions: Biological: IMA 401 (Phase Ib)

INTERVENTIONS:
Biological: IMA401 (Phase Ia) — Intravenous infusions in escalating dose levels
  Arms: Dose-Finding Combination Therapy with IMA401 TCER® and Pembrolizumab (Phase Ia); Dose-Finding IMA401 TCER® Monotherapy (Phase Ia)
Biological: Pembrolizumab (Phase Ia) — Intravenous infusions in escalating dose levels for combination of IMA 401 and Pembrolizumab
  Other Names: Keytruda®
  Arms: Dose-Finding Combination Therapy with IMA401 TCER® and Pembrolizumab (Phase Ia)
Biological: IMA 401 (Phase Ib) — Treatment at recommended dose for extension (RDE)
  Arms: Extension IMA401 TCER® Monotherapy (Phase Ib)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and initial anti-tumor activity of IMA401 as monotherapy or in combination with checkpoint inhibitor in patients with recurrent and/or refractory solid tumors.

Patients' HLA status and expression of the MAGE-A4 and/or MAGE-A8 target in the tumor must be confirmed.

Primary objective:

* To determine the maximum tolerated dose and/or recommended dose for extension for IMA401 as monotherapy and in combination with pembrolizumab

Secondary objectives:

* To characterize the safety and tolerability of IMA401 as monotherapy and in combination with pembrolizumab
* To evaluate initial anti-tumor activity of IMA401 as monotherapy and in combination with pembrolizumab
* To describe the pharmacokinetics of IMA401 as monotherapy and in combination with pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Patients must have voluntarily signed a written ICF, be able to understand and comply with clinical trial procedures
* Patients ≥ 18 years old
* Patients must have pathologically confirmed and documented advanced and/or metastatic NSCLC or HNSCC, other solid tumor may be considered
* Confirmed HLA status and IMA401 tumor target MAGE-A4 and/or MAGE-A8 expression
* Life expectancy > 2 months
* ECOG Performance Status of 0 to 1
* Measurable disease according to RECIST 1.1
* Adequate baseline hematologic, renal and hepatic function; acceptable coagulation status
* Patients must have recurrent and/or refractory solid tumors and must have received or not be eligible for all available indicated standard of care treatments
* The patient must have recovered from any side effects of prior therapy to Grade 1 or lower (except for non-clinically significant toxicities; e.g., alopecia, vitiligo) prior to treatment start. As determined by the investigator, the patient may still be eligible if the patient has not fully recovered from Grade ≥ 2 toxicities, in case if these toxicities are not anticipated to further improve (e.g., chronic peripheral neuropathy) and such toxicities are not anticipated to worsen with the IMA401 therapy

Exclusion Criteria:

* Other active malignancies that require treatment or that might interfere with the trial endpoints (ongoing adjuvant anti-hormonal treatment is allowed)
* History of hypersensitivity to components of IMA401, CPI treatment or rescue medications, contraindication for pembrolizumab
* Patients with prior allogeneic stem cell transplantation or organ transplantation
* Patients with autoimmune diseases needing disease-directed treatment
* Any serious or uncontrolled health condition, which, in the opinion of the Investigator, would place the subject at undue risk from the study, impair the ability of the subject to receive protocol specified therapy, or interfere with the interpretation of study results
* Positive for HIV or with active hepatitis B or C infection.
* Patients with active infection
* Systemic corticosteroids (≥ 10 mg/day prednisone or equivalent) received 2 weeks prior to starting trial treatment
* Patients with active central nervous system metastases and leptomeningeal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | 44 months

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) | 93 months
Number of patients with serious TEAEs | 93 months
Number of patients with treatment emergent adverse events of special interest (AESIs) | 93 months
Frequency of dose interruptions and reductions | 93 months
Duration of dose interruptions and reductions | 93 months
Overall response rate (ORR) based on best overall response (BOR) of complete response (CR) and partial response (PR) locally assessed using RECIST v1.1 and iRECIST | 93 months
Disease control rate (DCR) of CR, PR or stable disease (SD) lasting 6 or more weeks following the initiation of IMA401 | 93 months
Duration of response (DOR) of CR or PR based on RECIST v1.1 and iRECIST | 93 months
Progression-free survival (PFS) based on RECIST v1.1 and iRECIST | 93 months
Overall survival (OS) | 93 months
Determination of IMA 401 PK parameter: maximal serum concentration (Cmax) | 44 months
Determination of IMA 401 PK parameter: time at Cmax (Tmax) | 44 months
Determination of IMA 401 PK parameter: minimal serum concentration (Cmin) | 44 months
Determination of IMA 401 PK parameter: area under the serum concentration-time curve (AUC) | 44 months
Determination of IMA 401 PK parameter: clearance (Cl) | 44 months
Determination of IMA 401 PK parameter: volume of distribution (Vss) | 44 months
Determination of IMA 401 PK parameter: half-life (t1/2) | 44 months
Determination of IMA 401 PK parameter: assessment of dose-proportionality | 44 months
Determination of IMA 401 PK parameter: steady-state attainment | 44 months

CONTACTS AND LOCATIONS:
Overall Officials: Immatics Biotechnologies GmbH, Study Director — Immatics Biotechnologies GmbH
Locations (23):
- Germany (23):
  - Universitaetsklinikum Freiburg, Zentralklinikum, Klinik fuer Innere Medizin I, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg AöR, Nationales Zentrum fuer Tumorkrankheiten, Heidelberg, Baden-Wurttemberg
  - Thoraxklinik Heidelberg gGmbH, Studienzentrum Thoraxonkologie, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen AöR, Comprehensive Cancer Center Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm AöR, ECTU-Early clinical Trials Unit Universitaetsklinikum Ulm Comprehensive Cancer Center Ulm_CCCU, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen AöR, Interdisciplinary Clinical Trial Unit with ECTU, Erlangen, Bavaria
  - Klinikum rechts der Isar der TU Muenchen AöR, Klinik und Poliklinik fuer Innere Medizin III, Munich, Bavaria
  - Klinikum Nuernberg, Klinik fuer Innere Medizin 5, Abteilung Onkologie/Haematologie, Nuremberg, Bavaria
  - Universitaetsklinikum Regensburg AöR, Klinik fuer Innere Medizin 3, Regensburg, Bavaria
  - Universitaetsklinikum Wuerzburg AöR, Interdisziplinaeres Studienzentrum mit ECTU, Würzburg, Bavaria
  - Goethe Universitaetsklinikum Frankfurt AöR, Medizinische Klinik II, Frankfurt am Main, Hesse
  - Sana Klinikum Offenbach GmbH, Klinik für Pneumologie/ Thoraxzentrum Rhein-Main, Offenbach, Hesse
  - Universitätsmedizin Göttingen, Klinik für Hämatologie und Onkologie, Göttingen, Lower Saxony
  - Medizinische Hochschule Hannover, Klinik fuer Haematologie, Haemostaseologie, Onkologie und Stammzelltransplantation, Hanover, Lower Saxony
  - Universitätsklinikum Bonn AöR, Medizinische Klinik IIII, Bonn, North Rhine-Westphalia
  - Marien Hospital Duesseldorf GmbH, Klinik fuer Onkologie/Haematologie und Palliativmedizin, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Muenster AöR, Medizinische Klinik A, Münster, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, III. Medizinische Klinik, Mainz, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH, Klinik für Innere Medizin III, Chemnitz, Saxony
  - Universitaetsklinikum C. - G. - Carus Dresden, Technische Universitaet Dresden AöR, NCT/UCC Early Clinical Trial Unit, Dresden, Saxony
  - Universitaet Leipzig, Universitaeres Krebszentrum Leipzig (UCCL), Leipzig, Saxony
  - Universitaetsklinikum Schleswig- Holstein, Campus Kiel, Medizinische Klinik II Haematologie und Onkologie, Karl-Lennert Tumorzentrum, Kiel, Schleswig-Holstein
  - Charité Universitaetsmedizin Berlin KöR, Klinik fuer Haematologie und Onkologie, Berlin

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- See also: Corporate Website — http://immatics.com/